CLINICAL TRIAL: NCT02124694
Title: Iwankapiya-Healing: Historical Trauma Practice and Group IPT for American Indians
Acronym: HTUG-IPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R34MH097834-01A1 (NIH)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2016-05

CONDITIONS: Depression; Grief; PTSD; Interpersonal Relations
Keywords: historical trauma and unresolved grief; complicated grief; prolonged grief; interpersonal conflicts; depression; American Indians; interpersonal psychotherapy; traumatic grief; posttraumatic stress disorder
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Historical Trauma; Prolonged Grief Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HTUG and IPT (Experimental): This arm includes the Historical Trauma and Unresolved Grief intervention (HUTG) combined with group Interpersonal Psychotherapy (IPT).The HTUG/IPT arm is 12 two-hour sessions delivered weekly on average, except for weather delays, over 16 weeks. HTUG/IPT includes sessions on identifying relationship issues which may trigger depressive symptoms, using group support, and connecting the impact of collective tribal trauma and losses with personal lifespan and current losses. HTUG/IPT is aimed at reducing depressive symptoms related to interpersonal conflicts and grief. HTUG is a Tribal Best Practice which may serve to engage AI in IPT, an empirically supported treatment for depression.
  Interventions: Behavioral: HTUG
- IPT Only (No Intervention): IPT is a standard empirically supported treatment. This IPT Only group is not receiving the experimental HTUG component and is being compared to the combined HTUG with IPT.

INTERVENTIONS:
Behavioral: HTUG — HTUG is a group psychotherapy...
  Other Names: Historical Trauma and Unresolved Grief Intervention
  Arms: HTUG and IPT

SUMMARY:
This study will pilot an intervention that combines group Interpersonal Psychotherapy (IPT), an empirically-supported treatment, and the Historical Trauma and Unresolved Grief Intervention (HTUG), a Tribal Best Practice for American Indians. HTUG focuses on grief, depression, and trauma response resolution related to collective massive group trauma across generations, including the lifespan, for American Indians. We anticipate more positive responses to, and patient engagement in, the combined HTUG/IPT intervention than to IPT Only.

DETAILED DESCRIPTION:
In this pilot study (R34), we will explore the feasibility, acceptance and sustainability of a treatment engagement and retention strategy that combines the Historical Trauma and Unresolved Grief Tribal Best Practice (HTUG) and Group Interpersonal Psychotherapy (IPT). HTUG is designed to engage and retain American Indian (AI) adults in treatment by focusing on grief resolution related to AI collective massive group trauma across generations. The model has potential for engaging AIs in empirically supported or evidence based treatments (EBTs) through the acknowledgment of the negative effects of colonialism on well-being and reducing the stigma of mental health problems. This study will test HTUG's potential to engage AIs in IPT, an EBT that may be particularly well suited for treating depression and related mental disorders in this population. IPT has demonstrated efficacy for treatment of depression and grief in diverse populations, and promising results to date with PTSD; however, to our knowledge, IPT has not been studied with AIs.

The specific aims for this proposal are:

1. Manualize, field test, and refine a combined group HTUG/IPT intervention model and related clinician training and research protocols. Under Aim 1, we will: a) develop HTUG/IPT model and initial manual, b) refine IPT for use with AIs, c) solicit AI Advisory Panel (AP) member and clinician review of models, d) prepare pilot measures, e) prepare HTUG/IPT training materials, and f) recruit and train providers.
2. Conduct a pilot randomized trial of HTUG/IPT compared to IPT Only at two sites (Albuquerque, New Mexico and Pine Ridge Indian Reservation, South Dakota) to further refine the manual and protocols, and assess the feasibility and acceptability of our procedures for conducting a subsequent large-scale clinical trial. Under Aim 2, we will conduct the randomized trial in two waves; we will: a) recruit participants, b) implement interventions and collect data, c) analyze data, and d) develop "products" - the finalized HTUG/IPT manual, an R01 proposal, conference presentations and manuscripts, and the final manual and data report to the two clinics.

Upon completion of these aims, we will have piloted methods and established the feasibility and acceptance of the HTUG/IPT intervention model, which will provide foundational data for an R01 to test strategies for improving engagement and retention of AIs in EBTs. What is learned in the proposed program of research could have significant promise for reducing disparities in mental health treatment and disease burden across AI populations and in culturally unique, disadvantaged and poorly served populations in general. Improving engagement and retention in culturally relevant EBTs among AIs is of great practical importance given the rates of lifetime prevalence of mental health disorders (ranging from 35% to 54%), the fact that mental health care for AIs is severely underfunded, and the reality that treatment research with AIs is sorely lacking.

Two sites are participating in this project in two different Indian Health Service (IHS) Areas: Southwest urban and Northern Plains reservation outpatient behavioral health clinics. These include First Nations Community HealthSource in the Albuquerque Area in New Mexico and Oglala Lakota College/Kyle Health Center on the Pine Ridge Reservation in the Aberdeen Area in South Dakota. Participants will be randomly assigned to either the IPT Only treatment or the combined HTUG/IPT group; both will be 12 two hour sessions of group intervention. We anticipate that the HTUG/IPT group will show increased positive response to the intervention as measured on a number of scales for depression, grief, and interpersonal functioning as well as satisfaction with the model. We will use the results to design a more in-depth randomized clinical trial (R01) at additional tribal sites.

ELIGIBILITY:
Inclusion Criteria

* American Indian adults
* Depression
* Co-occurring unresolved, prolonged or complicated grief included
* Co-occurring PTSD or other trauma response included
* Score of 16 on Hamilton Depression Scale and clinician assessment
* DSM 5 Substance Use Disorder Mild for alcohol or cannabis only or remission

Exclusion Criteria:

* Psychosis
* Personality disorder
* Bipolar disorder
* Severe vegetative depressive symptoms such as psychomotor retardation
* Acutely suicidal or homicidal individuals
* Mild, moderate or severe substance abuse disorder for amphetamines, methamphetamines, opioids, hallucinogens or inhalants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-04-22 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Changes in Hamilton Depression Scale from Baseline | Initial Screening, two mid-points (weeks 4 and 8), end of intervention (week 12) and follow up (8 weeks post intervention)
  Scale commonly used in IPT studies to assess depressive symptoms and track change over time. The Ham -D24 (and other shorter versions) is a commonly used clinician-administered depression assessment scale. This HAM-D24 is a 24 item version that incorporates three new items that assess helplessness, hopelessness, and worthlessness. The measure is commonly used to rate the severity of, and change in, a patient's major depression. It includes 24 items rated on a scale from 0-2, 0-3, or 0-4, with a total score computed ranging from 0-75. An earlier version of the Hamilton Depression Rating Scale the HAM-D17 has the following psychometric properties: Cronbach's alphas have been found to range from 0.46 to 0.97; inter-rater reliability, Pearson's r ranged from 0.82 to 0.98; and the intraclass r ranged from 0.46 to 0.99. The HAM-D24 is believed to have similar psychometric properties.

SECONDARY OUTCOMES:
Changes in the PCL PTSD Checklist | Initial Screening, two mid-points (weeks 4 and 8), end of intervention (week 12) and follow up (8 weeks post intervention)
  The PCL is a 17-item self-report measure of the 17 DSM-IV symptoms of PTSD. The PCL is used to screening individuals for PTSD, diagnosing PTSD, and monitoring symptom change during and after treatment. A total symptom severity score (range = 17-85) can be obtained by summing the scores from each of the 17 items. The PCL has good internal consistency, with a Cronbach's alpha of .86.
Changes on the Historical Losses and Historical Losses Associated Symptoms Scales (HLS/HLAS) | Baseline, end of intervention (12 weeks), and 8 weeks follow up post-intervention
  Historical Losses and Historical Losses Associated Symptoms Scales - The items selected for HLS were determined by a series of focus groups conducted with elders in two tribes in the upper Midwest to identify the kinds of losses associated with historical trauma and the types of emotions felt when thinking about those losses. The HLAS asks how often the respondent feels each of 12 symptoms (e.g. anger, sadness, like the loss is happening again) when they think about the losses. The scale has good internal reliability, with a Cronbach's alpha of .89.
Changes in the Inventory of Complicated Grief (ICG) | Baseline, end of intervention (12 weeks), and 8 weeks follow up post-intervention
  The ICG assesses indicators of pathological grief, such as anger, disbelief, and hallucinations. It consists of 19 first-person statements concerning the immediate bereavement-related thoughts and behaviors of the client, with 5 response options ranging from "Never" to "Always." The ICG's internal consistency is good, with a Cronbach's alpha of .94. The test-retest reliability has been found to be .80. The scale has a well validated clinical cut point, with individuals scoring over 25 considered at risk for requiring clinical care.
Inventory of Interpersonal Problems (IIP) | Baseline, end of intervention (12 weeks), and 8 weeks follow up post-intervention
  The IIP is a self-report measure that identifies an individual's most salient interpersonal difficulties. There are two forms: The IIP-64 contains 64 statements describing common interpersonal problems. Scales include: Domineering/ Controlling, Vindictive/Self-Centered, Cold/Distant, Socially Inhibited, Nonassertive, Overly Accommodating, Self-Sacrificing, and Intrusive/Needy. Respondents rate how distressed they have been by each problem on a scale from 0 (not at all) to 4 (extremely). The IIP scales have adequate internal consistency and test-retest reliability.
Duke-UNC Functional Support Questionnaire | Baseline, end of intervention (12 weeks), and 8 weeks follow up post-intervention
  This questionnaire measures social support, which can be related to depression.
Medication Adherence Questionnaire | baseline, two mid-points (Week 4 and 8), end of intervetion and 8 week follow up
  this questionnaire was developed for implementation with research participants to assist in tracking the compliance with any current medication management that the participant is currently engaging in with their primary health care or behavioral health care provider. This is to see if the current medications are appropriate and helpful with depressive symptoms being experienced by the participant prior to entering into the study and during their participation in the study. This is part of Treatment as Usual to which research participants are entitled and is part of good clinical care.
Group Environment Scale | Two mid points (Weeks 4 and 8)
  Developed by Moos, Insel, and Humphrey this measure is to assess group climate and comfort level of the study participants to openly discuss issues related to the target symptoms of depression in group. Clinical group facilitators/staff at each study site will complete the observational measure.
Group Engagement Measure | Two mid points (Weeks 4 and 8)
  is a comprehensive measure to assess the various dimensions of group engagement by study participants. This will be completed by research team members

OTHER OUTCOMES:
Indigenous Peoples Survey (IPS) | Baseline
  The IPS is a clinician administered instrument for collective group trauma, lifetime trauma exposure, tribal cultural identity values and practices, religiosity/spirituality and the experiencing of racism and discrimination on mental health symptoms and associated outcomes. The IPS is an investigator constructed measure grounded in prior work on HTUG. The IPS includes questions about tribal cultural identity, values and practices; health and mental health; grief, trauma exposure and symptoms; and experiences of racism and discrimination. It includes investigator constructed questions and standardized measures, with the intent that AI mental health clinics could use the IPS to conduct more comprehensive assessments framed in a culturally resonant structure.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Y Brave Heart, PhD, Principal Investigator — University of New Mexico Department of Psychiatry
Locations (1):
- University of New Mexico Department of Psychiatry Center for Rural and Community Behavioral Health, Albuquerque, New Mexico, United States